CLINICAL TRIAL: NCT07120815
Title: Optimizing Metformin Use in Polycystic Ovary Syndrome - A Randomized Controlled Trial
Brief Title: Optimizing Metformin Use in Polycystic Ovary Syndrome
Acronym: MET-PCOS
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Valtion tutkimusraha (funding) (Unknown); Sakari Alhopuro foundation (funding) (Unknown); The Medical Society of Finland (funding) (Unknown)
Responsible Party: Principal Investigator, Johanna Melin, MD, PhD, specialist in obstetrics & gynecology, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HUS8428/TYH2024323; 2023-509259-15-01 (EU CTIS Number)
Record Dates: First submitted 2025-07-09; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Polycystic Ovary Syndrome (PCOS)
Keywords: polycystic ovary syndrome; metformin; randomized controlled trial
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Women 18-37 years old with a BMI ≥ 25 kg/m2, metformin 2250mg per day (Active Comparator): metformin tablets 2250 mg per day
  Interventions: Drug: Metformin 2250 mg daily
- Women 18-37 years old with a BMI ≥ 25 kg/m2, metformin 1500mg per day (Experimental): metformin tablets 1500 mg per day
  Interventions: Drug: Metformin 1500 mg daily

INTERVENTIONS:
Drug: Metformin 1500 mg daily — metformin 500mg tablets, 3 times per day
  Arms: Women 18-37 years old with a BMI ≥ 25 kg/m2, metformin 1500mg per day
Drug: Metformin 2250 mg daily — Metformin 750mg, 3 times daily
  Arms: Women 18-37 years old with a BMI ≥ 25 kg/m2, metformin 2250mg per day

SUMMARY:
The goal of this clinical trial is to learn if a metformin dose of 1500 mg or 2250 mg per day is better to treat polycystic ovary syndrome (PCOS) in adults. It will also learn about the adverse effects of metformin. The trial aims to evaluate which metformin dose is better for:

1. improving biochemical and clinical outcomes
2. gastrointestinal side-effects
3. mental health and quality of life

Participants will:

* Be randomized to take metformin at a dose of either 1500mg or 2250mg every day for 6 months
* Visit the clinic three times during the trial for checkups and tests
* Answer questionnaires on menstrual cyclicity, mental health, quality of life and side-effects

DETAILED DESCRIPTION:
INTRODUCTION Polycystic ovary syndrome (PCOS) remains a key public health burden as it is one of the most common endocrine and metabolic disorders affecting up to 13% of women globally. The Rotterdam diagnostic criteria were updated and internationally endorsed in the 2023 International PCOS guideline and include a) ovulatory and menstrual dysfunction, b) biochemical and/or clinical hyperandrogenism and c) polycystic ovary morphology (PCOM) at ultra-sound. For a diagnosis in adults two of three criteria are required, with PCOM remaining nonspecific for PCOS in adolescents.

Women with PCOS present with diverse features; metabolic (weight gain, obesity, insulin resistance and diabetes) reproductive (infertility and pregnancy complications), endocrine (hyperandrogenism, hirsutism and acne) and psychosocial (depression, anxiety and poor quality of life).

While lifestyle management is strongly recommended for weight management, for those with higher body mass index (BMI), sustainable efficacy for weight loss can be limited and additional pharmacological treatment may be needed. The 2023 Updated International PCOS Guideline recommends that metformin, in addition to lifestyle, should be considered in adults with PCOS and BMI ≥ 25 kg/m2 for prevention of weight gain and management of weight and metabolic disorders. Metformin may be considered in adults with BMI < 25 kg/m2 and adolescents with PCOS, acknowledging more limited evidence.

The aim of this randomized controlled trial (RCT) is to evaluate whether a metformin dose of 1500 mg is inferior compared to a dose of 2250 mg per day for females 18-37 years of age with PCOS in:

1. improving biochemical and clinical outcomes
2. gastrointestinal side-effects
3. mental health and quality of life

MATERIALS AND METHODS A double-blind, randomized controlled trial, including adults (age 18-37 years) with PCOS and a BMI ≥ 25 kg/m2 will be carried out. The randomization will be computer-generated and performed by the hospital pharmacy with 1:1 allocation in random blocks. Power analysis has indicated that a total number of 184 females (92 in each group) will be needed to reveal a 4 kg weight reduction (equals 5% weight reduction for a person weighting 80 kg) with an 80% power. We estimated a 15% drop-out in our power analysis.

Potential participants for the study will be recruited from females referred to the Reproductive Medicine Unit at Helsinki University Hospital and by advertising via the patient organization for those with PCOS (Korento). The internationally indorsed Rotterdam criteria will be used to diagnose women with PCOS. Pregnant women, women breastfeeding, women with untreated thyroid disease, hyperprolactinemia, other conditions with hyperandrogenism or use of hormonal contraceptive during the last three months will be excluded.

Women willing to participate in the study will be randomized to metformin 1500mg or 2250 mg per day for a 6-month period. Blood samples (on hyperandrogenism and metabolism), clinical examination (anthropometry and hirsutism) and a questionnaire (menstrual cyclicity, mental health, quality of life, side-effects) will be performed before starting the metformin medication, as well as at 3 and 6 months after onset of medication. Polycystic ovary morphology will be evaluated by measuring anti-mullerian hormone levels (AMH) and by vaginal ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed PCOS (According to the International evidence-based Guideline for PCOS 2023)
* Age: 18-37 years
* BMI: ≥ 25 and <40 kg/m2
* Signed informed consent and willingness to comply with the trial procedures
* Sufficient skills in the Finnish or Swedish language

Exclusion Criteria:

* Not meeting the criteria according to the International evidence-based Guideline for PCOS 2023)
* Use of hormonal contraceptive during the last 3 months
* Pregnancy
* Breastfeeding
* Untreated diabetes
* Hypothyroidism
* Hyperprolactinemia
* Use of medications for diabetes,
* Use of medications for high cholesterol
* Use of medications for obesity
* Use of medications for cortisone (per oral)
* Hypersensitivity to metformin
* Acute metabolic acidosis
* Renal impairment
* Hepatic insufficiency
* Heart- or respiratory failure
* Serious mental illness
* Alcoholism
* Investigator site staff directly involved in the conduct of the study and their family members

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 184 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Weight | The investigators will measure change in outcomes from baseline to 14 and 26 weeks
  Weight will be measured by a standard scale to an accuracy of +/- 0,1kg.
Homeostatic model assessment for insulin resistance (HOMA-IR) | The investigators will measure change in outcomes from baseline to 14 and 26 weeks
  HOMA-IR will be calculated with the formula: fasting plasma glucose (mmol/L) × fasting serum insulin (mU/L) divided by 22.5 (9)
Hirsutism | The investigators will report change from baseline to 14 and 26 weeks.
  Modified Ferriman Gallwey score (mFG) will be measured and a score of 4 or more will be regarded as hirsutism in Caucasian women, whereas a score of 6 or more will be regarded hirsutism for other ethnicities
Total testosterone | The investigators will measure change from baseline to 14 and 26 weeks
  Testosterone nmol/l (liquid chromatography with tandem mass spectrometry (LC-MS/MS). All laboratory tests will be taken in the morning, between 7-10 am, after 12 hours fasting.
Appearance of severe of adverse effects | The investigators will measure change from baseline to 14 and 26 weeks
  In our questionnaire the investigators will ask the participants whether they have experienced abdominal pain, reflux, nausea, diarrhoea or loss of appetite during the last two weeks and grade the symptoms from 1-5 (1 being never and 5 being all the time). The investigators will count the scores and give each participant a score between 5-25. A severe adverse effect is defined as a score of 4 or more in one of the questions (indicating a daily experience of abdominal pain, reflux, nausea, diarrhoea or loss of appetite during the last two weeks).
Anti-Mullerian hormone (AMH) | The investigators will measure change from baseline to 14 and 26 weeks
  AMH will be measured in ug/l. All laboratory tests will be taken in the morning, between 7-10 am, after 12 hours fasting.

SECONDARY OUTCOMES:
Body mass index (BMI) | The investigators will measure change in outcomes from baseline to 14 and 26 weeks
  Weight (kilogram) and height (metre) will be combined to report BMI in kg/m^2
Waist circumference (WC) | The investigators will measure change in outcomes from baseline to 14 and 26 weeks
  WC will be measured halfway between the participant's lowest rib and the top of the participant's hipbone
Waist-hip-ratio (WHR) | The investigators will measure change in outcomes from baseline to 14 and 26 weeks
  WHR will be calculated as waist measurement divided by hip measurement (W⁄H). Hip circumference is determined as the maximum value over the glottal region, measured to the nearest centimetre.
Body adiposity index (BAI) | The investigators will measure change in outcomes from baseline to 14 and 26 weeks
  BAI will be measured using the following equation: hip circumference (cm)/height (m) - 18
Body composition | The investigators will measure change in outcomes from baseline to 14 and 26 weeks
  Body composition will be measured with a multi-frequency segmental body composition analyzer (TANITA Health Ware) WHR (Waist-hip-ratio). Will be calculated as waist measurement divided by hip measurement (W⁄H). Hip circumference is determined as the maximum value over the glottal region, measured to the nearest centimetre.
  WC (Waist circumference). Measured halfway between the participant's lowest rib and the top of the participant's hipbone BAI (Body adiposity index). Will be measured using the following equation: hip circumference (cm)/height (m) - 18 BP (blood pressure) (systolic and diastolic) and pulse. Will be measured twice with at least 3 minutes apart after at least 10 min rest from non-dominant upper extremity in a subject in supine position
Blood pressure (BP) | The investigators will measure change in outcomes from baseline to 14 and 26 weeks
  BP (systolic and diastolic) will be measured twice with at least 3 minutes apart after at least 10 min rest from non-dominant upper extremity in a subject in supine position
Pulse | The investigators will measure change in outcomes from baseline to 14 and 26 weeks
  Pulse will be measured twice with at least 3 minutes apart after at least 10 min rest from non-dominant upper extremity in a subject in supine position
Fasting glucose | The investigators will measure change in outcomes from baseline to 14 and 26 weeks
  fasting glucose mmol/l (photometric hexokinase method) All laboratory tests will be taken in the morning, between 7-10 am, after 12 hours fasting.
Fasting insulin | The investigators will measure change in outcomes from baseline to 14 and 26 weeks
  fasting insulin mU/l (immunochemiluminometric assay) All laboratory tests will be taken in the morning, between 7-10 am, after 12 hours fasting.
HbA1C | The investigators will measure change in outcomes from baseline to 14 and 26 weeks
  HbA1C mmol/mol (photometric enzymatic method) All laboratory tests will be taken in the morning, between 7-10 am, after 12 hours fasting.
Lipids (cholesterol and its subclasses, triglycerides) | The investigators will measure change in outcomes from baseline to 14 and 26 weeks
  Total cholesterol, mmol/l and triglycerides mmol/l with an enzymatic photometric method, LDL and HDL mmol/l with a direct enzymatic photometric method All laboratory tests will be taken in the morning, between 7-10 am, after 12 hours fasting.
C-reactive protein (CRP) | The investigators will measure change in outcomes from baseline to 14 and 26 weeks
  CRP will be measured in mg/l (photometric immunochemical method) All laboratory tests will be taken in the morning, between 7-10 am, after 12 hours fasting.
2-hour oral glucose tolerance test (OGTT) | The investigators will measure change in outcomes from baseline to 14 and 26 weeks
  2-hour OGTT mmol/l
Alanine Aminotransferase (ALAT) | The investigators will measure change in outcomes from baseline to 14 and 26 weeks
  ALAT will be measured in U/l (photometric method according to the International Federation of Clinical Chemistry and Laboratory Medicine recommendation) All laboratory tests will be taken in the morning, between 7-10 am, after 12 hours fasting.
Gamma-glutamyl transferase (G-GT) | The investigators will measure change in outcomes from baseline to 14 and 26 weeks
  G-GT will be measured in U/l (photometric method according to the International Federation of Clinical Chemistry and Laboratory Medicine recommendation) All laboratory tests will be taken in the morning, between 7-10 am, after 12 hours fasting.
Fatty Liver Index (FLI) | The investigators will measure change in outcomes from baseline to 14 and 26 weeks
  FLI will be measured by the following formula:
  FLI = (e^y) / (1 + e^y) * 100 where: y = 0.953 * ln(TG) + 0.139 * BMI + 0.718 * ln(GGT) + 0.053 * WC - 15.745 e is the base of the natural logarithm (approximately 2.718) ln denotes the natural logarithm TG is triglycerides in mg/dL BMI is body mass index in kg/m² GGT is gamma-glutamyltransferase in U/L WC is waist circumference in cm All laboratory tests will be taken in the morning, between 7-10 am, after 12 hours fasting.
Matsuda Index | The investigators will measure change in outcomes from baseline to 14 and 26 weeks
  Matsuda Index will be measured by the following formula:
  Matsuda Index = 10,000 / √[(fasting glucose (mg/dL) * fasting insulin (µU/mL)) * (mean glucose (mg/dL) * mean insulin (µU/mL) during OGTT) All laboratory tests will be taken in the morning, between 7-10 am, after 12 hours fasting.
Triglyceride-Glucose (TyG) index | The investigators will measure change in outcomes from baseline to 14 and 26 weeks
  TyG Index will be measured by the following formula:
  TyG Index=fasting triglycerides (mg/dL) * fasting glucose (mg/dL) / 2 All laboratory tests will be taken in the morning, between 7-10 am, after 12 hours fasting.
Acne | The investigators will report change from baseline to 14 and 26 weeks
  The investigators will use the PCOS-Q to ask about acne (score 1-7)
Alopecia | The investigators will report change from baseline to 14 and 26 weeks
  The investigators will use the PCOS-Q to ask about alopecia (score 1-7)
Free androgen index (FAI) | The investigators will measure change from baseline to 14 and 26 weeks
  FAI will be calculated with the following formula:
  FAI = 100 X ((Total Testosterone (nmol/L)/SHBG (nmol/L)) All laboratory tests will be taken in the morning, between 7-10 am, after 12 hours fasting.
Sex hormone binding globulin (SHBG) | The investigators will measure change from baseline to 14 and 26 weeks
  SHBG will be measured in nmol/l (immunochemiluminometric assay) All laboratory tests will be taken in the morning, between 7-10 am, after 12 hours fasting.
Dehydroepiandrosterone sulfate (DHEAS) | The investigators will measure change from baseline to 14 and 26 weeks
  DHEAS will be measured in nmol/l (immunochemiluminometric assay) All laboratory tests will be taken in the morning, between 7-10 am, after 12 hours fasting.
Androstenedione | The investigators will measure change from baseline to 14 and 26 weeks
  Androstenedione will be measured in nmol/l (liquid chromatography with tandem mass spectrometry (LC-MS/MS) All laboratory tests will be taken in the morning, between 7-10 am, after 12 hours fasting.
Free testosterone | The investigators will measure change from baseline to 14 and 26 weeks
  Free calculated testosterone will be measured in pmol/l (by Anderson Formula). All laboratory tests will be taken in the morning, between 7-10 am, after 12 hours fasting.
Menstrual regularity | The investigators will measure change from baseline to 14 and 26 weeks
  Questionnaire, where asking if the menstrual cycle is regular (defined as 21 days or more but under 36 days)
Menstrual cycle length | The investigators will measure change from baseline to 14 and 26 weeks
  Questionnaire, where asking how long the two previous cycles were (days)
Appearance of gastrointestinal adverse effects (GI AE) | The investigators will measure change from baseline to 14 and 26 weeks
  In our questionnaire the investigators will ask the participants whether they have experienced abdominal pain, reflux, nausea, diarrhoea or loss of appetite during the last two weeks and grade the symptoms from 1-5 (1 being never and 5 being all the time). The investigators will count the scores and give each participant a score between 5-25. A severe adverse effect is defined as a score of 4 or more in one of the questions (indicating a daily experience of abdominal pain, reflux, nausea, diarrhoea or loss of appetite during the last two weeks).
Quality of life (QoL) | The investigators will measure change from baseline to 14 and 26 weeks
  The PCOS-Q is a questionnaire that was specifically designed to measure quality of life for women with PCOS. Questions on depression, anxiety, fear etc will be given scores from 1-7, depending on severity.
Weight stigma | The investigators will measure change from baseline to 14 and 26 weeks
  In the questionnaire appearance of weight stigma and examples on it will be asked.
Follicle number per ovary (FNPO) and antral follicle count (AFC) | The investigators will measure change from baseline to 14 and 26 weeks.
  Vaginal ultrasound where the investigators measure FNPO and AFC will be performed at any stage of the cycle.
Ovarian volume | The investigators will measure change from baseline to 14 and 26 weeks.
  Vaginal ultrasound where the investigators measure ovarian volume will be performed at any stage of the cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Johanna M Melin, MD, Principal Investigator — The Reproductive Medicine Unit, Helsinki University Hospital
Locations (1):
- The Reproductive Medicine Unit, Helsinki University Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant-level data, including demographic information, medical history, laboratory results, and outcome data, will be shared. A data dictionary detailing variable names and coding will also be provided.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available starting 6 months after publication and remain accessible for 2 years.
Access Criteria: Access will be granted to qualified researchers with a valid research proposal and a signed data sharing agreement. Data will be anonymized to protect participant privacy. Informed consent procedures will be reviewed to ensure participants were aware of data sharing practices.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-15): https://cdn.clinicaltrials.gov/large-docs/15/NCT07120815/Prot_SAP_000.pdf